CLINICAL TRIAL: NCT03669731
Title: Evaluation of the Protein Intake of the Pregnant Woman According to the Weight Status and in Pregnant Women Operated on Bariatric Surgery
Acronym: BariaProG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CHU-405; 2017-A02350-53 (Other: 2017-A02350-53)
Record Dates: First submitted 2018-08-30; First posted 2018-09-13 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Pregnant Women From 20 Amenorrhea Weeks
Keywords: Obesity; Protein; Pregnancy; bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Diet Records

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Urinary urea 24 hours and food diary
  Interventions: Other: food diary
- Group 2 (Experimental): Urinary urea 24 hours and food diary
  Interventions: Other: food diary
- Group 3 (Experimental): Urinary urea 24 hours and food diary
  Interventions: Other: food diary

INTERVENTIONS:
Other: food diary — This food diary is to be completed by the patient in the 3rd trimester of pregnancy, on 3 consecutive days and if possible including a weekend day. Finally, the investigator also prescribes a biological analysis: a urinary urea from a 24h diuresis to be collected in the 3rd trimester in a dedicated collector and given that same day.

SUMMARY:
Adequate equipment for lifelong health is essential to ensure healthy health for fetal development. In France, pregnant women with normal weight have increased protein intake to 0.78-0.95g / kg / day (ANC 2001). And more recently, AFSSA from 2007 proposed a recommended nutritional intake of 0.82-1g / kg / d. An increased requirements in the second and third trimester of 0.25 g / kg / day and 0.46 g / kg / day, respectively, compared with non-pregnancy values. However, the prevalence of the incompatibility remains unknown.

In addition, maternal protein intake is inadequate or excessively associated with both intra-uterine growth retardation and small gestational age weights. Neonatal hypotrophy is also associated with a risk of chronic diseases in adulthood, including cardiovascular disease, type 2 diabetes, insulin resistance, high blood pressure and coronary heart disease.

In obese women or patients undergoing surgery for bariatric surgery, there is currently no recommendation on the recommended protein intake. Or, maternal obesity plays a role in the metabolic development of children and bariatric surgery is associated with a major risk of maternal micronutrient deficiencies and intra-uterine growth retardation.

Prevalence of obesity in France is currently estimated at 17%. Moreover, bariatric surgery is also fast-growing in France with a number of interventions having tripled since 2006.

Thus, a better understanding of maternal food needs and applications throughout pregnancy is needed to improve dietary guidelines and promote fetal, neonatal and long-term health.

DETAILED DESCRIPTION:
The main objective is to evaluate the protein intake of the pregnant woman in the 3rd trimester of pregnancy in 3 populations:

* Women with BMI ≥ 18.5 and <30 kg / m² (group 1)
* Obese women (BMI ≥ 30 kg / m²) (group 2)
* Women operated on a bariatric surgery (group 3)

ELIGIBILITY:
Inclusion Criteria:

* - Pregnant women from 20 amenorrhea weeks.
* Women aged at least 18 years old.
* Women with BMI ≥ 18.5 and <30 kg / m² = Group 1
* Obese women (BMI ≥ 30 kg / m²) = Group 2
* Women operated on a bariatric surgery (by-pass, sleeve-gastrectomy, gastric band) = Group 3

Exclusion Criteria:

* - Women with BMI <18.5 kg / m²
* Troubles of eating behavior
* Women with gestational diabetes
* Medical history of type 1 or type 2 diabetes
* Multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Protein intake | an average of 33 weeks
  In the 3rd trimester = Weight adjusted protein intake (g / kg / day) ± total protein intake (g / d) and protein proportion of total caloric intake (%) using a 3-day diary.

SECONDARY OUTCOMES:
link between protein consumption in the 3rd trimester and ultrasound data | an average of 33 weeks
  For the 3 groups: results of all obstetrical ultrasound exams performed at 20 AS
nutritional state (nutritional deficiencies) of pregnant women operated on a bariatric surgery using the biological results at T1, T2, T3. | an average of 7,20 and 33 weeks
  Retrospective collection of the results of the biological assessment prescribed in the three trimesters (including vitamins, trace elements) for the group of women operated on bariatric surgery
protein requirements of the pregnant woman according to the 3 groups | an average of 33 weeks
  The protein requirement of the patients is determined from a statistical analysis called straight line of linear regression between nitrogen balance and protein intake (g / kg / day body weight) for the population. It corresponds, according to this line, to the value for which the nitrogen balance is zero.

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France